CLINICAL TRIAL: NCT04186416
Title: Effectiveness of the Pressure Recording Analytical Method in Predicting the Fluid Responsiveness in Pediatric Surgical Critical Care Patients
Brief Title: Effectiveness of the Pressure Recording Analytical Method in Predicting Fluid Responsiveness in Pediatric Critical Care Patients
Acronym: MOSTCARE-PED
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191036; 2019-A02804-53 (Other: IDRCB number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hypovolemia; Hemorrhage; Fluid Responsiveness
Keywords: Volume expansion in children; Mostcare® device; Fluid responsiveness; Stroke volume; Transthoracic cardiac echocardiography
MeSH Terms: conditions — Hypovolemia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients less than 6 months old: Patients less than 6 months old admitted to the pediatric surgical ICU of the Necker-Enfants Malades university hospital and for whom volume expansion is indicated.
  Interventions: Other: Mostcare® device; Other: Transthoracic cardiac ultrasound
- Patients between 6 and 12 months old: Patients between 6 and 12 months old admitted to the pediatric surgical ICU of the Necker-Enfants Malades university hospital and for whom volume expansion is indicated.
  Interventions: Other: Mostcare® device; Other: Transthoracic cardiac ultrasound
- Patients between 1 and 6 years old: Patients between 1 and 6 years old admitted to the pediatric surgical ICU of the Necker-Enfants Malades university hospital and for whom volume expansion is indicated.
  Interventions: Other: Mostcare® device; Other: Transthoracic cardiac ultrasound
- Patients between 6 and 10 years old: Patients between 6 and 10 years old admitted to the pediatric surgical ICU of the Necker-Enfants Malades university hospital and for whom volume expansion is indicated.
  Interventions: Other: Mostcare® device; Other: Transthoracic cardiac ultrasound

INTERVENTIONS:
Other: Mostcare® device — The Moscare® system is connected to the patient monitoring devices. Data are collected just before and 5 minutes after the vascular filling.
Other: Transthoracic cardiac ultrasound — Transthoracic cardiac ultrasound before and 3 minutes after the vascular filling.

SUMMARY:
The Pressure Recording Analytical Method, invasive hemodynamic monitoring, is an uncalibrated pulse contour analysis, installed in the Mostcare® system that allows a continuous estimation of the stroke volume and thus the cardiac output, by the relationship between the area under the curve of the systolic portion of the arterial blood pressure curve and the dynamic impedance of the cardiovascular system.

The objectives of the study are to determine if the parameters measured by Mostcare® make it possible to predict the response to volume expansion in pediatric surgical critical care patients, sedated, intubated and ventilated, by comparing the changes in stroke volume, induced by a volume expansion, measured by trans-thoracic echocardiography.

DETAILED DESCRIPTION:
Children undergoing major surgery or severe trauma with bleeding require regular hemodynamic evaluation, including cardiac output measurement, to maintain adequate organ perfusion. In fact, administration of fluid to improve cardiac output is the mainstay of hemodynamic resuscitation. However, not all patients respond to fluid therapy, and excessive fluid administration is harmful. Therefore, the vascular filling strategy requires a thorough hemodynamic evaluation.

Many predictive tools for fluid responsiveness have been validated in adults, and are based on heart-lung interaction in ventilated patients. Up to now, respiratory variation in aortic blood flow peak velocity, measured by transthoracic or transoesophageal cardiac echocardiography, is the only variable shown to effectively predict fluid responsiveness in children.

However, the use of these methods does not allow continuous monitoring (trans-thoracic echocardiography) or is not easily achievable in current practice (trans-esophageal echocardiography). In addition, these monitoring tools require learning and inter- and intra-individual variability is not negligible, ranging from 1% to 20%.

The Pressure Recording Analytical Method, invasive hemodynamic monitoring, is an uncalibrated pulse contour analysis, installed in the Mostcare® system, that allows a continuous estimation of the stroke volume and thus of the cardiac output, by the relationship between the area under the curve of the systolic portion of the arterial blood pressure curve and the dynamic impedance of the cardiovascular system.

The goal of this study is to assess the ability of dynamic cardiovascular variables measured using Mostcare® to predict fluid responsiveness in pediatric surgical critical care patients, sedated, intubated and ventilated, in prone position, by comparing the changes in stroke volume (SV), induced by a volume expansion (VE), measured by trans-thoracic echocardiography. For the purpose of the study, responders (Rs) to VE are patients showing an increase in SV measured using transthoracic echocardiography of at least 15% after VE.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 10 years old, of both sexes.
* Perioperative period of surgery under general anesthesia requiring admission to surgical resuscitation (before and / or after the surgical procedure).
* Patients admitted for severe trauma.
* Patient installation: supine position.
* Intubation and mechanical ventilation: tidal volume: 7 to 8 ml / kg, Positive expiratory pressure : 3-4 cm H2O, inspiration / expiration: 1 / 1.5 to 1/2; respiratory rate: 1 month up to 2 years = 30 / min; children 2-8 years = 20 / min; children> 8 years = 15 / min.
* Patients with arterial catheters.
* Need for a volume expansion : indication given by the doctor in charge of the patient.
* Non-opposition expressed by the holders of parental authority.

Exclusion Criteria:

* Cardiac rhythm disorders (in particular atrial fibrillation, junctional tachycardia, ventricular arrhythmias), with the exception of sinus tachycardia, respiratory variations of heart rate and sporadic atrial / ventricular extrasystoles whom will allow inclusion.
* Cardiopathy: severe systolic dysfunction (shortening fraction <28%, ejection fraction <50%); valvulopathy (significant narrowing or valvular insufficiency); left-right shunt, persistent arterial duct.
* Unstable hemodynamic status related to active bleeding requiring vascular filling > 2 mL / kg / min or requiring vasopressor or inotropic therapy whose dosage had to be changed in the last five minutes.
* Need for mechanical ventilation with a tidal volume> 10 mL / kg or <7 mL / kg.
* Refusal of the patient or the holders of parental authority to exploit the collected data.
* Impossibility to carry out measurements.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients between birth and 10 years of age admitted to the pediatric surgical ICU of the Necker-Enfants Malades university hospital and for whom volume expansion is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Stroke volume variation from Mostcare® | 5 minutes after infusion of bolus fluid
  Predictability of stroke volume variation (SVV) from Mostcare® for fluid responsiveness.
  Patients are defined as responders if stroke volume obtained using echocardiography increased by ≥15% after volume expansion.

SECONDARY OUTCOMES:
Absolute values and variation of cardiac output (CO) and cardiac index (CI) from Mostcare® | 5 minutes after infusion of bolus fluid
  Correlation with CO and CI measured by transthoracic cardiac ultrasound before and after volume expansion.
Absolute values and variation of stroke volume (SV) and indexed stroke volume (SVi) from Mostcare® | 5 minutes after infusion of bolus fluid
  Correlation with SV and SVi by transthoracic cardiac ultrasound before and after volume expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Orliaguet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Estelle Vergnaud, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No